CLINICAL TRIAL: NCT06394336
Title: Efficacy of an Early Intervention Programme Using Therapeutic Exercise in Patients With Plantar Fasciopathy
Brief Title: Early Intervention With Therapeutic Exercise in Plantar Fasciopathy
Acronym: PIPex-FP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Javier Marco Lledó, Universidad Miguel Hernández, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ProtocoloFP
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Plantar Fascitis
Keywords: therapeutic exercise; strengthening

STUDY DESIGN:
Intervention Model Description: Experimental study with random allocation of patients with similar characteristics to the control and intervention groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): People with PF who will receive the usual treatment (oral analgesic/anti-inflammatory drug) prescribed by the primary care physician and will also participate in the therapeutic exercise programme.
  Interventions: Other: Muscle strengthening
- Non-experimental group (Active Comparator): Individuals with PF who will receive the usual treatment (oral analgesic/anti-inflammatory drug) prescribed by the primary care physician
  Interventions: Drug: Standard treatment (oral analgesic/anti-inflammatory drug)

INTERVENTIONS:
Other: Muscle strengthening — Strengthening exercises for the intrinsic muscles of the foot and hips
  Arms: Experimental group
Drug: Standard treatment (oral analgesic/anti-inflammatory drug) — oral analgesic/anti-inflammatory drug. Education.
  Arms: Non-experimental group

SUMMARY:
The aim of this project is to evaluate the efficacy of a therapeutic exercise programme in patients with plantar fasciitis applied early and aimed at strengthening the hip and foot musculature.

DETAILED DESCRIPTION:
All patients will be informed about the study to be carried out and will give their prior informed consent. The programme has a first part of teaching directed to patients by physiotherapists, and a second part of application at home, with a duration of 12 weeks. An experimental study will be designed with random assignment of patients with similar characteristics to two groups. The non-experimental group will receive their usual treatment (medication and recommnendations as stretching) and the experimental group will follow their usual treatment and also participate in the therapeutic programe.

ELIGIBILITY:
Inclusion Criteria:

* Patients with referred pain in the medial plantar area of the heel, accentuated with initial steps after a period of inactivity but also worsening after prolonged body weight bearing, of at least 3 months evolution prior to inclusion in the study.
* Reproduction of the pain referred by the patient with palpation at the proximal insertion of the plantar fascia.

Exclusion Criteria:

* Pregnancy.
* Injection of corticoids in the area in the 6 months prior to recruitment.
* Previous illnesses that may alter gait (central or peripheral neurological pathology, degenerative and inflammatory arthropathies, systemic illnesses).
* Existence of concomitant foot pathology (metatarsalgia, stress fractures, neuropathies due to entrapment, tendinitis, history of foot/ankle surgery, etc.).
* People who do not have the capacity to understand and follow an exercise programme.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2024-05-10 (Estimated); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | It will be assessed at baseline and at 12 weeks (at the end of the intervention period), with a subsequent follow-up period at 3 and 6 months after the end of the intervention.
  For its estimation a numerical pain rating scale will be used, where 0 represents no pain (at all) and 10, the worst pain imaginable. Using this instrument the patient should rate the intensity of pain at the start of walking in the morning (the first step), the worst time of the day and the average level of pain the participant has experienced in the last week. This is an easy to complete, quick and simple scale. A 2-point change on this scale is a clinically important difference in people with chronic pain.
Disability | It will be assessed at baseline and at 12 weeks (at the end of the intervention period), with a subsequent follow-up period at 3 and 6 months after the end of the intervention.
  To be estimated using the Spanish version of the foot function index. The FFI consists of 23 items divided into 3 subscales that quantify the impact of foot pathology on pain, disability and activity limitation.
General health and health-related quality of life: | It will be assessed at baseline and at 12 weeks (at the end of the intervention period), with a subsequent follow-up period at 3 and 6 months after the end of the intervention.
  Is a generic instrument for measuring health-related quality of life. It has 5 health dimensions: mobility, self-care, activities of daily living, pain/discomfort and anxiety/depression. Each of these has three levels of severity
Physical activity | It will be assessed at baseline and at 12 weeks (at the end of the intervention period), with a subsequent follow-up period at 3 and 6 months after the end of the intervention.
  t will be measured through the International Physical Activity Questionnaire (IPAQ). This questionnaire consists of 7 items. The aim of this instrument is to record the degree of physical activity, sitting hours and walking time of the subjects who complete it.
Overall perception of clinical change | It will be assessed at baseline and at 12 weeks (at the end of the intervention period), with a subsequent follow-up period at 3 and 6 months after the end of the intervention.
  The overall rating of change will be obtained using an 11-point scale. It measures the overall perceived change in the condition of their heel pain from the time they started the study to the present as "worse", "no change" or "better".

CONTACTS AND LOCATIONS:
Overall Officials: Javier Marco, PhD, Study Chair — Universidad Miguel Hernandez de Elche
Locations (1):
- Hospital General Universitario de Elche, Elche, Alicante, Spain

REFERENCES:
- [Background] Buchanan BK, Sina RE, Kushner D. Plantar Fasciitis. 2024 Jan 7. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK431073/ PMID 28613727
- [Background] Budiman-Mak E, Conrad KJ, Mazza J, Stuck RM. A review of the foot function index and the foot function index - revised. J Foot Ankle Res. 2013 Feb 1;6(1):5. doi: 10.1186/1757-1146-6-5. PMID 23369667
- [Background] Cheung RT, Sze LK, Mok NW, Ng GY. Intrinsic foot muscle volume in experienced runners with and without chronic plantar fasciitis. J Sci Med Sport. 2016 Sep;19(9):713-5. doi: 10.1016/j.jsams.2015.11.004. Epub 2015 Nov 22. PMID 26655866
- [Background] Goff JD, Crawford R. Diagnosis and treatment of plantar fasciitis. Am Fam Physician. 2011 Sep 15;84(6):676-82. PMID 21916393
- [Background] Kamonseki DH, Goncalves GA, Yi LC, Junior IL. Effect of stretching with and without muscle strengthening exercises for the foot and hip in patients with plantar fasciitis: A randomized controlled single-blind clinical trial. Man Ther. 2016 Jun;23:76-82. doi: 10.1016/j.math.2015.10.006. Epub 2015 Oct 30. PMID 26654252
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Latey PJ, Burns J, Hiller CE, Nightingale EJ. Relationship between foot pain, muscle strength and size: a systematic review. Physiotherapy. 2017 Mar;103(1):13-20. doi: 10.1016/j.physio.2016.07.006. Epub 2016 Aug 4. PMID 27986277
- [Background] Lim AT, How CH, Tan B. Management of plantar fasciitis in the outpatient setting. Singapore Med J. 2016 Apr;57(4):168-70; quiz 171. doi: 10.11622/smedj.2016069. PMID 27075037
- [Background] Luffy L, Grosel J, Thomas R, So E. Plantar fasciitis: A review of treatments. JAAPA. 2018 Jan;31(1):20-24. doi: 10.1097/01.JAA.0000527695.76041.99. PMID 29227320
- [Background] Pascual Huerta J. The effect of the gastrocnemius on the plantar fascia. Foot Ankle Clin. 2014 Dec;19(4):701-18. doi: 10.1016/j.fcl.2014.08.011. Epub 2014 Sep 26. PMID 25456717
- [Background] Spink MJ, Fotoohabadi MR, Menz HB. Foot and ankle strength assessment using hand-held dynamometry: reliability and age-related differences. Gerontology. 2010;56(6):525-32. doi: 10.1159/000264655. Epub 2009 Dec 3. PMID 19955706
- [Background] Sullivan J, Burns J, Adams R, Pappas E, Crosbie J. Musculoskeletal and activity-related factors associated with plantar heel pain. Foot Ankle Int. 2015 Jan;36(1):37-45. doi: 10.1177/1071100714551021. Epub 2014 Sep 18. PMID 25237175
- [Background] Sullivan J, Pappas E, Burns J. Role of mechanical factors in the clinical presentation of plantar heel pain: Implications for management. Foot (Edinb). 2020 Mar;42:101636. doi: 10.1016/j.foot.2019.08.007. Epub 2019 Sep 3. PMID 31731071
- [Background] Yoo SD, Kim HS, Lee JH, Yun DH, Kim DH, Chon J, Lee SA, Han YJ, Soh YS, Kim Y, Han S, Lee W, Han YR. Biomechanical Parameters in Plantar Fasciitis Measured by Gait Analysis System With Pressure Sensor. Ann Rehabil Med. 2017 Dec;41(6):979-989. doi: 10.5535/arm.2017.41.6.979. Epub 2017 Dec 28. PMID 29354574
- [Background] Rathleff MS, Molgaard CM, Fredberg U, Kaalund S, Andersen KB, Jensen TT, Aaskov S, Olesen JL. High-load strength training improves outcome in patients with plantar fasciitis: A randomized controlled trial with 12-month follow-up. Scand J Med Sci Sports. 2015 Jun;25(3):e292-300. doi: 10.1111/sms.12313. Epub 2014 Aug 21. PMID 25145882
- [Background] Riel H, Vicenzino B, Jensen MB, Olesen JL, Holden S, Rathleff MS. The effect of isometric exercise on pain in individuals with plantar fasciopathy: A randomized crossover trial. Scand J Med Sci Sports. 2018 Dec;28(12):2643-2650. doi: 10.1111/sms.13296. Epub 2018 Oct 1. PMID 30203866
- [Background] Franettovich Smith MM, Collins NJ, Mellor R, Grimaldi A, Elliott J, Hoggarth M, Weber Ii KA, Vicenzino B. Foot exercise plus education versus wait and see for the treatment of plantar heel pain (FEET trial): a protocol for a feasibility study. J Foot Ankle Res. 2020 May 8;13(1):20. doi: 10.1186/s13047-020-00384-1. PMID 32384905